CLINICAL TRIAL: NCT02524158
Title: Yoga Therapy to Improve Function Among Veterans With Chronic Low Back Pain
Brief Title: Yoga for Veterans With CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O7768-R
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Chronic Low Back Pain
Keywords: Yoga; Mind-Body Therapies; Chronic Low Back Pain; Military Veterans; VA patients
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): The yoga intervention will consist of 2x weekly, 60-minute Hatha Yoga classes for 12 weeks, geared toward a CLBP population. Classes begin with a few minutes of simple seated breathing exercises. Depending on their mobility, participants can sit either on the floor or on a chair. This is followed by gentle warm-up stretches. Participants are then led through a series of standing postures, seated postures and floor postures. The difficulty of the poses will gradually increase over the duration of the 12 weeks, and appropriate modifications are offered to participants whenever needed. Deep and rhythmic breathing will be emphasized throughout. Each class will end with a supine resting pose.
  Interventions: Behavioral: Yoga Therapy for CLBP
- Delayed Treatment Control - Usual Care (No Intervention): Participants randomly assigned to this arm are allowed to continue all existing treatments. Participants and their primary care physician are asked to not change treatments unless medically necessary. participants are asked to not do yoga for 6 months. They are given free yoga and a yoga mat after 6 months.

INTERVENTIONS:
Behavioral: Yoga Therapy for CLBP — Classes begin with a few minutes of simple seated breathing exercises. Depending on their mobility, participants can sit either on the floor or on a chair. This is followed by gentle warm-up stretches. Participants are then led through a series of standing postures, seated postures and floor postures. The difficulty of the poses will gradually increase over the duration of the 12 weeks, and appropriate modifications are offered to participants whenever needed. Deep and rhythmic breathing will be emphasized throughout. Each class will end with a supine resting pose.
  Arms: Yoga

SUMMARY:
Chronic low back pain (CLBP) is a prevalent condition among VA patients, but many current treatment options have limited effectiveness. In addition to chronic pain, people with chronic low back pain experience increased disability, psychological symptoms such as depression, and reduced health-related quality of life. This randomized controlled study will examine the impact of yoga therapy for improving function and decreasing pain in VA patients with chronic low back pain. Although not every VA patient with chronic low back pain will choose to do yoga, it is an inexpensive treatment modality that is increasingly appealing to many VA patients. If yoga is effective, it could become an additional low-cost option that the VA can offer to better serve Veterans with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Has a VA primary care provider
* Diagnosis of chronic low back pain > 6 months
* Willing to attend a yoga program or be assigned to delayed treatment with yoga
* Willing to complete 4 assessments
* English Literacy
* Has not begun new pain treatments or medications in the past month
* Willing to not change pain treatments (e.g., discontinue a treatment; increase medication dose) during the 12-week intervention period unless medically necessary

Exclusion Criteria:

* back surgery within the last 12 months
* back pain due to specific systemic problem (eg, lupus, scleroderma, fibromyalgia)
* morbid obesity (BMI > 40)
* Significant sciatica or nerve compression < 3 months or chronic lumbar radicular pain > 3 months
* Unstable, serious coexisting medical illness (eg, CHF, cancer, COPD, morbid obesity; dementia)
* Unstable, serious psychiatric illness (e.g., unmanaged psychosis, active substance dependence)
* Insufficient data to rule out acute, metastatic disease, (unless primary care physician approves)
* Attended or practiced yoga > 1x in the last 12 months
* Positive Romberg test (with or without sensory neuropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik J Groessl, PhD BA BS, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groessl EJ, Liu L, Richard EL, Tally SR. Cost-effectiveness of Yoga for Chronic Low Back Pain in Veterans. Med Care. 2020 Sep;58 Suppl 2 9S:S142-S148. doi: 10.1097/MLR.0000000000001356. PMID 32826784
- [Derived] Groessl EJ, Liu L, Chang DG, Wetherell JL, Bormann JE, Atkinson JH, Baxi S, Schmalzl L. Yoga for Military Veterans with Chronic Low Back Pain: A Randomized Clinical Trial. Am J Prev Med. 2017 Nov;53(5):599-608. doi: 10.1016/j.amepre.2017.05.019. Epub 2017 Jul 20. PMID 28735778

RESULTS

PARTICIPANT FLOW:
Groups:
- Yoga: The yoga intervention consisted of 2x weekly, 60-minute Hatha Yoga classes for 12 weeks. Classes begin with a few minutes of simple seated breathing exercises. Depending on their mobility, participants can sit either on the floor or on a chair. This is followed by gentle warm-up stretches. Participants are then led through a series of standing postures, seated postures and floor postures. The difficulty of the poses will gradually increase over the duration of the 12 weeks, and appropriate modifications are offered to participants whenever needed. Deep and rhythmic breathing will be emphasized throughout. Each class will end with a supine resting pose.
Period: 12-weeks Assessment
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Started | 76 | 76
Completed | 57 | 63
Not Completed | 19 | 13
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 18 | 12
Period: 6-month Assessment
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Started | 76 | 76
Completed | 54 | 55
Not Completed | 22 | 21
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 21 | 20

BASELINE CHARACTERISTICS:
Population: Of the 76 participants randomized to each group, 1 participants in each group requested withdrawal of all of their data from the study. Thus, baseline characteristics, outcomes analyses, and outcomes results are reported for 75 participants.
Groups:
- Yoga: The yoga intervention consisted of 2x weekly, 60-minute Hatha Yoga classes for 12 weeks, geared toward a CLBP population. Classes begin with a few minutes of simple seated breathing exercises. Depending on their mobility, participants can sit either on the floor or on a chair. This is followed by gentle warm-up stretches. Participants are then led through a series of standing postures, seated postures and floor postures. The difficulty of the poses will gradually increase over the duration of the 12 weeks, and appropriate modifications are offered to participants whenever needed. Deep and rhythmic breathing will be emphasized throughout. Each class will end with a supine resting pose.
- Total: Total of all reporting groups
Arm/Group | Yoga | Delayed Treatment Control - Usual Care | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.7) | 53.6 (13.9) | 53.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 55 | 56 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 60 | 60 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 10 | 26
  White | 50 | 54 | 104
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Roland-Morris Disability Questionnaire
Description: The primary outcomes is the change in Roland-Morris Disability Questionnaire (RMDQ) score between baseline and 12-weeks. The questionnaire consists of 24 questions that ask about back pain-related functional limitations experienced for a variety of daily activities . Scores can range from 0-24. Higher scores indicate more impairment, and when considering the change from baseline to follow-up assessments, negative scores indicate improvement. The scale has been shown to be reliable and is well validated. It has been used in another yoga RCT, allowing for comparisons.
Time Frame: baseline to 12 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 75 | 75
units on a scale | -2.05 [-3.18 to 0.92] | -1.29 [-2.36 to -0.22]
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.340, Mixed Models Analysis

2. Primary Outcome: Roland-Morris Disability Questionnaire
Description: The primary outcome is the change in Roland-Morris Disability Questionnaire (RMDQ) score between baseline, 12-weeks, and 6-months. The questionnaire consists of 24 questions that ask about back pain-related functional limitations experienced for a variety of daily activities . Scores can range from 0-24. Higher scores indicate more impairment, and when considering the change from baseline to follow-up assessments, negative scores indicate improvement. The scale has been shown to be reliable and is well validated. It has been used in another yoga RCT, allowing for comparisons.
Time Frame: baseline to 6-months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 75 | 75
units on a scale | -3.37 [-4.51 to -2.23] | -0.89 [-2.02 to 0.23]
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.003, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline in Pain Intensity - Brief Pain Inventory at 12 Weeks
Description: The short version of the Brief Pain Inventory (BPI) is a self-rated questionnaire designed to assess the severity of pain and the impact of pain on daily functions in the past day and week. The BPI takes about 5 minutes to complete and has been validated with low back pain patients. It has been shown to respond to both behavioral and pharmacological pain interventions. The BPI measures severity of pain, impact of pain on daily function, location of pain, pain medications, and amount of pain relief. Items are answered utilizing a scoring algorithm, with the mean of the 4 severity items used as measures of pain severity. Scores range from 0-10, with higher scores indicating more pain, and when considering the change from baseline to follow-up assessments, negative scores indicate improvement.
Time Frame: baseline to 12 weeks
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 75 | 75
units on a scale | -0.61 [-0.94 to -0.28] | 0.04 [-0.27 to 0.35]
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.005, Mixed Models Analysis — The a priori specified threshold is p < 0.05

4. Secondary Outcome: Change From Baseline in Pain Intensity - Brief Pain Inventory at 6 Months
Description: as for outcome 3
Time Frame: baseline to 6 months
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 75 | 75
units on a scale | -0.44 [-0.78 to -0.11] | 0.15 [-0.18 to 0.47]
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.013, Mixed Models Analysis

5. Secondary Outcome: Change From Baseline Pain Interference - Brief Pain Inventory at 12 Weeks
Description: The short version of the Brief Pain Inventory (BPI) is a self-rated questionnaire designed to assess the severity of pain and the impact of pain on daily functions in the past day and week. The BPI takes about 5 minutes to complete and has been validated with low back pain patients. It has been shown to respond to both behavioral and pharmacological pain interventions. The BPI measures severity of pain, impact of pain on daily function, location of pain, pain medications, and amount of pain relief. Items are answered utilizing a scoring algorithm, with the mean of the 7 interference items used a as a measure of pain interference. Scores range from 0-10, with higher scores indicating more pain, and when considering the change from baseline to follow-up assessments, negative scores indicate improvement.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Yoga: The yoga intervention will consist of 2x weekly, 60-minute Hatha Yoga classes for 12 weeks, geared toward a CLBP population.
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 75 | 75
units on a scale | -0.85 (0.245) | -0.21 (0.217)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.044, ANCOVA — The a priori specified threshold is p < 0.05

6. Secondary Outcome: Change From Baseline - Fatigue Severity Scale (FSS) at 12 Weeks
Description: Fatigue (absence of energy) will be measured with the Fatigue Severity Scale (FSS). The FSS is a self-administered instrument developed to assess the impact and severity of fatigue. It consists of 9 items describing the functional impact of fatigue on daily life rated on a scale from 1 (strongly disagree) to 7 (strongly agree) with the total fatigue score ranging from 9-63 or an average score ranging from 1.0-7.0. Higher scores reflect greater fatigue severity and less energy.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 57 | 62
units on a scale | -5.29 (1.532) | 0.82 (1.172)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p < 0.01, ANCOVA

7. Secondary Outcome: Change From Baseline - SF12 PCS at 12 Weeks
Description: Health-related quality of life will be measured using the Short-form 12 (SF12). Based on the longer SF-36, the SF-12 was developed with the objective of finding a short yet meaningful measure of generic HRQOL or global health status. The 12 items were selected from the SF-36 and tested through a series of stages. The PCS-12 and MCS-12 show similar levels of precision to the summary scores derived from the longer 36-item measure. PCS-12 and MCS-12 scores are transformed to a 0 to 100, with higher scores indicating better quality of life.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 57 | 63
units on a scale | 4.40 (1.042) | 0.58 (0.853)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.010, ANCOVA — The a priori specified threshold is p < 0.05

8. Secondary Outcome: Change From Baseline - SF12 MCS at 12 Weeks
Description: Mental Component Scale - Health-related quality of life will be measured using the Short-form 12 (SF12). Based on the longer SF-36, the SF-12 was developed with the objective of finding a short yet meaningful measure of generic HRQOL or global health status. The 12 items were selected from the SF-36 and tested through a series of stages. The PCS-12 and MCS-12 show similar levels of precision to the summary scores derived from the longer 36-item measure. PCS-12 and MCS-12 scores are transformed to a 0 to 100, with higher scores indicating better quality of life.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 57 | 63
units on a scale | -0.04 (1.024) | -0.43 (0.772)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.66, ANCOVA

9. Secondary Outcome: Change From Baseline - EuroQOL 5D (EQ5D) at 12 Weeks
Description: The EQ5D is a preference-based measure of health-related quality of life. The measure produces a single score ranging from 0 (death) to 1.00 (optimal health). Scores can be integrated with time to calculate Quality Adjusted Life Years.
Time Frame: baseline to 12 weeks
Population: Main outcomes were conducted using linear modeling across multiple time points. This analysis used only 2 time points, with attrition from the 12-week assessment, and incomplete answers accounting for reduced sample size.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 59 | 61
units on a scale | 0.077 [0.031 to 0.122] | 0.018 [-0.023 to 0.060]
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p < 0.10, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline - Center for Epidemiologic Studies Short Depression Scale (CES-D 10) at 12 Weeks
Description: Depression will be assessed using the Center for Epidemiologic Studies Short Depression Scale (CES-D 10). Derived from the full CES-D, there are 10 items that ask about the frequency of mood symptoms, rated on a 4-point Likert scale ranging from 0 (Never) to 3 (All of the Time). Scores range from 0 to 30, and higher scores indicate greater depression. A number of items are reverse-scored and a score of 10 or greater is considered depressed. Normative data on people with assorted chronic illnesses are available for comparisons.
Time Frame: baseline to 12 weeks
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 56 | 62
units on a scale | -1.6 (0.549) | -0.63 (0.499)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.202, ANCOVA

11. Secondary Outcome: Change From Baseline - Brief Anxiety Inventory (BAI) at 12 Weeks
Description: The Brief Anxiety Inventory (BAI) measures the severity of anxiety symptoms, particularly those that distinguish anxiety from depression. The BAI consists of 21 items, is self-administered and can be completed in 5 to 10 minutes. Items are scored on a scale of 0 to 3 and are summed to generate a total score. Scores range from 0 to 63, and higher scores indicate greater depression.
Time Frame: baseline to 12 weeks
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 55 | 55
units on a scale | -1.69 (1.08) | 0.23 (0.67)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.369, ANCOVA

12. Secondary Outcome: Change From Baseline - Pittsburgh Sleep Quality Index (PSQI) at 12 Weeks
Description: The PSQI is a validated measure of sleep quality. The global PSQI score has a range of 0-21, with higher scores indicating worse sleep quality.
Time Frame: baseline to 12 weeks
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 55 | 61
units on a scale | -1.56 (0.43) | -0.082 (0.41)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.50, ANCOVA

13. Secondary Outcome: Change From Baseline - Self-efficacy for Managing Low Back Pain at 12 Weeks
Description: Self-efficacy for controlling CLBP reflects levels of confidence in the ability to influence the intensity of back pain symptoms and the impact that CLBP has on daily life. The questions are based on self-efficacy items developed for the Medical Outcomes Study in mixed chronic diseases. The wording of the items has been adapted to be specific to CLBP. The measure consists of 6 items, rated on a 6-point Likert scale, with each item ranging from 0-10. The total score is the mean of the 6 items with higher scores indicating greater self-efficacy for managing CLBP.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 57 | 63
units on a scale | 0.26 (0.27) | -0.48 (0.21)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.067, ANCOVA

14. Secondary Outcome: Attendance/ Home Practice
Description: Two indicators of the amount of yoga practiced by each participant will be used. Actual attendance of yoga sessions will be assessed using VA medical record data. Attendance can range from 0-24 sessions attended for those participants randomized to yoga. Self-reported practice of yoga at home will be assessed using a weekly participant yoga log. The self-report yoga log assesses whether they practiced yoga each day, the amount of minutes practiced, the use of instructions, the difficulty of poses, and the estimated level of physical activity or exertion.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: sessions attended
Groups:
- Yoga: Participants randomized at baseline to receive 2x weekly yoga for 12 weeks.
Arm/Group | Yoga
Number analyzed (Participants) | 75
sessions attended | 12.28 (1.013)

15. Secondary Outcome: Change From Baseline - Range of Motion - Flexion at 12 Weeks
Description: Spinal Range of Motion (ROM) will be measured using a Saunders Digital Inclinometer, a portable device which isolates lumbar ROM. The device is placed along the spine and uses a precise optical angular scanner. Forward bend angle measures how far forward and downward a person can bend at the waist, from a fully erect and/or normal standing position. The value typically ranges from 0-180 degrees, with higher values indicating greater flexibility.
Time Frame: baseline to 12 weeks
Population: Only a subset agreed to assessment. Some declined if concerned about injury. Main outcomes were conducted using linear modeling across multiple time points. This analysis used only 2 time points, with attrition from the 12-week assessment, and incomplete answers accounting for reduced sample size.
Measure: Mean (Standard Error); unit: degrees flexion
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 44 | 49
degrees flexion | 7.41 (2.56) | 2.65 (2.24)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.071, ANCOVA

16. Secondary Outcome: Change From Baseline - Grip Strength at 12 Weeks
Description: Grip strength in both hands of each participant will be measured using an adjustable, hydraulic grip strength dynamometer (Jamar Hydraulic Hand Dynamometer). Three trials will be conducted for each hand. In cases of current pain flare-ups or recent procedures to a hand or wrist, the affected hand is not tested, and the result of the one other hand is used. If both hands are used the best performance of two trials will be selected for each side, and the average of the left and right hand will be used for analysis. The value measured is pounds of force exerted and typically ranges from 0 - 150 lbs, with higher numbers indicating greater grip strength.
Time Frame: baseline to 12 weeks
Population: Some participants declined to participate because of injury concern. Main outcomes were conducted using linear modeling across multiple time points. This analysis used only 2 time points, with attrition from the 12-week assessment, and incomplete answers accounting for reduced sample size.
Measure: Mean (Standard Error); unit: pounds per sq inch
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 42 | 49
pounds per sq inch | -0.30 (1.59) | 0.62 (1.17)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.92, ANCOVA

17. Secondary Outcome: Change From Baseline - Lower Limb Strength and Balance - Eyes Open at 12 Weeks
Description: The Single Leg Stance (SLS) is a commonly used measure of both lower leg strength and balance. A total of four trials were conducted - left and right leg with both eyes open and eyes closed. Each trial will be timed from the moment the participant lifts one foot off the floor until the moment they need to place it on the floor again. If the participant is able to stand on one leg for 60 seconds the trial will be stopped and they will be asked to switch side. Values range from 0 - 60 seconds with greater values indicating better balance.
Time Frame: baseline to 12 weeks
Population: as for outcome 15
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 43 | 49
seconds | 6.21 (2.63) | 1.05 (1.34)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.036, ANCOVA — The a priori specified threshold is p < 0.05

18. Secondary Outcome: Change From Baseline - Lower Spine Stabilization - Core Strength at 12 Weeks
Description: Time in seconds holding plank position on the elbows.
Time Frame: baseline to 12 weeks
Population: as for outcome 15
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
Number analyzed (Participants) | 40 | 44
seconds | 18.70 (4.15) | 10.50 (3.28)
Statistical Analysis 1: Comparison: Yoga vs Delayed Treatment Control - Usual Care; Test type: Superiority; p = 0.071, ANCOVA

ADVERSE EVENTS:
Arm/Group | Yoga | Delayed Treatment Control - Usual Care
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 2/75 | 0/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=75) | Delayed Treatment Control - Usual Care (N=75)
Increased back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — One participant reported increased levels of back pain after one session and declined to attend further. A second participant attended 7 consecutive yoga sessions and stopped attending because his "back went out" and pain increased.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No